CLINICAL TRIAL: NCT03730051
Title: Contrast Enhanced Breast MRI: Comparison of Two Macrocyclic Gadolinium-Based Contrast Agents: Gadoterate Meglumine (Dotarem) and Gadobutrol (Gadavist). A Prospective Study.
Brief Title: Dotarem vs Gadobutrol Contrast for Breast MRI
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Principal Investigator, Gopal Vijayaraghavan, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H00020209
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-03

CONDITIONS: Breast Diseases
Keywords: Breast MRI; Mammography; Dotarem contrast; Gadobutrol contrast; wash-in/wash-out contrast curve; Contrast enhanced MRI
MeSH Terms: conditions — Breast Diseases | interventions — gadoterate meglumine; gadobutrol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gadoterate meglumine contrast (Active Comparator): 0.2 mL/kg (0.1 mmol/kg) administered as a single IV bolus injection at a rate of 2 mL/second. The FDA-approved product labeling provides weight-adjusted dose volumes as follows: 30 kg: 6 mL; 40 kg: 8 mL; 50 kg: 10 mL; 60 kg: 12 mL; 70 kg: 14 mL; 80 kg: 16 mL; 90 kg: 18 mL; 100 kg: 20 mL; 110 kg: 22 mL; 120 kg: 24 mL; 130 kg: 26 mL; 140 kg: 28 mL; 150 kg: 30 mL.
  Interventions: Drug: Gadoterate meglumine
- Gadobutrol contrast (Experimental): 0.1 mL/kg (0.1 mmol/kg) administered as a single IV bolus injection by power injector. Imaging may begin after administration and then repeat sequentially to determine peak intensity and wash-out. The manufacturer provides weight-based dose volumes as follow: 35 kg: 3.5 mL; 40 kg: 4 mL; 45 kg: 4.5 mL; 50 kg: 5 mL; 60 kg: 6 mL; 70 kg: 7 mL; 80 kg: 8 mL; 90 kg: 9 mL; 100 kg: 10 mL; 110 kg: 11 mL; 120 kg: 12 mL; 130 kg: 13 mL; 140 kg: 14 mL.
  Interventions: Drug: Gadobutrol

INTERVENTIONS:
Drug: Gadoterate meglumine — Participants randomized into this arm will receive gadoterate meglumine contrast for their scheduled breast MRI.
  Other Names: Dotarem
  Arms: Gadoterate meglumine contrast
Drug: Gadobutrol — Participants randomized into this arm will receive gadobutrol contrast for their scheduled breast MRI.
  Other Names: Gadavist
  Arms: Gadobutrol contrast

SUMMARY:
In this randomized clinical trial, the investigators expect to demonstrate that the MRI contrast agent Dotarem is not less effective in contrast enhancement of breast lesions then Gadavist. Participants will be randomized to receive either Dotarem or Gadavist. In all cases, inclusion criteria will require patients having undergone or scheduled or most likely to be scheduled to undergo tissue sampling with histology results available. The patients will be prospectively and consecutively identified such that the majority of patients included will have been diagnosed with breast cancer, while including benign disease in the minority of patients in each arm. Following randomized enrollment, quantitative, semi-quantitative and qualitative image analysis will be performed to objectively assess for differences in image quality and diagnostic value.

DETAILED DESCRIPTION:
A stratified randomization of participants based on the time of menstural cycle and breast density. Women will then receive their clinically indicated Breast MRI with contrast, using SOC procedures for weight-based dosage. After enrollment, MRI images and medical metadata will be abstracted using the hospital medical records in EPIC and PACS databases. Data to be collected from the medical record includes histology parameters: tumor, tumor type and size, grade, stage and personal data: MRN, accession number, date of birth, date of MRI, age, sex, race/ethnicity, family history. Images will be stripped of identifiers and then coded by a study ID using the third party SanteSoft Dicom Editor software. Medidata will also be coded and stored separately from a mastercode file linking the study ID with the following identifiable information: MRN, accession number, date of birth, and date of MRI.

After a period of data collection, two radiologists blinded to the contrast agent will independently review the the MRIs. This qualitative review will consist of each exam being graded on a scale of 1-(Fail) to 5-(Excellent) contrast enhancement quality. Additionally, each blinded radiologist or designee will conduct the secondary quantitative measurements of the wash-in/wash-out contrast characteristics through use of computer aid design (CAD) in PACS.

ELIGIBILITY:
Inclusion Criteria:

* Females age 18 and older
* Scheduled to undergo a clinically indicated MRI of the breast with contrast.
* Have undergone, are scheduled to undergo, or are likely to be scheduled to undergo a breast tissue sampling exam with histology results available within 6 months of their MRI.

Exclusion Criteria:

* Pregnant
* Have already begun therapeutic treatment for breast cancer including surgery (lumpectomy or mastectomy), radiotherapy, or chemotherapy.
* Pre Menopause women outside of the 7-14 days from cycle

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 258 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of breast MRI | 6 months
  Each MRI exam will be graded by two radiologists blinded to the contrast agent using a scale of 1-(Fail- No enhancement or inadequate enhancement of the tumor) to 5-(Excellent- Strong and divisive contrast enhancement of entire tumor when compared to background. Clear and obvious tumor borders.) for the contrast enhancement quality.

SECONDARY OUTCOMES:
Wash-in/wash-out MRI contrast curve in breast tissues | 12 months
  The wash-in/wash-out MRI contrast curve will be assessed by software that analyzes the MRI images pixel by pixel for signal intensity changes over time on the breast MRI for each participant.
Maximum relative enhancement (E(max) for contrast breast MRI | 12 months
  The maximum relative enhancement (E(max)) will be assessed by software that analyzes the MRI images pixel by pixel for signal intensity changes over time on the breast MRI for each participant.
Time to peak enhancement (T(max)) for contrast breast MRI | 12 months
  The mean +/-sd of the time to peak enhancement (T(max)) will be assessed by software that analyzes the MRI images pixel by pixel for signal intensity changes over time on the breast MRI for each participant.
Maximum enhancement slope for contrast breast MRI | 12 months
  The maximum enhancement slope will be assessed by software that analyzes the MRI images pixel by pixel for signal intensity changes over time on the breast MRI for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Bloch, MD, Principal Investigator — UMASS Medical School
Locations (1):
- UMass Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No